CLINICAL TRIAL: NCT06892574
Title: A Trial of Rehabilitation Paired with VNS for Motor Function Recovery in Post-ICH Patients (Recovery Study)
Brief Title: Rehabilitation Paired with VNS for Motor Function Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, De-zhi Kang, Prof., First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 82371466
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Spontaneous Intracerebral Hemorrhage; Motor Function; Upper Extremity Injury; Rehabilitation; Vagus Nerve Stimulation
Keywords: Stroke; Hemorrhagic Stroke; Upper Extremity Paresis; Vagus Nerve Stimulation; Neuromodulation; Randomized Controlled Trial; Rehabilitation
MeSH Terms: conditions — Arm Injuries; Stroke; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The device can be set as active VNS or sham VNS (the actual intensity is 0 mA). An unmasking programmer not involved in treatments or assessments will be messaged the group of the participant and set appropriate stimulation setting at baseline follow-up timepoint. Other masking researchers, including therapists and assessors, as well as the participant will not know the stimulation setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VNS group (Experimental): Active VNS paired with rehabilitation Device: VNS A neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve.
  Other: Rehabilitation Rehabilitation movements to improve upper limb function after stroke.
  Interventions: Device: Active-VNS
- Control group (Sham Comparator): Sham VNS paired with rehabilitation Device: Sham VNS A neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve, the actual intensity is 0 mA.
  Other: Rehabilitation Rehabilitation movements to improve upper limb function after stroke.
  Interventions: Device: Sham VNS

INTERVENTIONS:
Device: Active-VNS — A neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve.
  Arms: VNS group
Device: Sham VNS — A neuromodulation treatment that delivers electrical impulses to the brain via the vagus nerve, the actual intensity is 0 mA.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of vagus nerve stimulation (VNS) combined with rehabilitation in improving upper extremity motor function after spontaneous intracerebral hemorrhage (ICH).

Researchers will evaluate the efficacy and safety of VNS by comparing the improvements of arm motor function post-ICH in the active VNS combined rehabilitation group with that in the sham VNS combined rehabilitation group (actual intensity 0 mA).

Participants in this study will undergo a surgical procedure to implant the VNS system and will subsequently recieve a 6 weeks in-clinic therapy, followed by an additional 6 weeks home exercise. During the final 6 weeks, participants will either recieve in-clinic therapy or maintain their home exercise, depending on their assigned group.

DETAILED DESCRIPTION:
There are 6 follow-up timepoints in this trial:

1. Screening follow-up timepoint (V1): All participants will sign the informed consent form and receive pre-implant evaluation, including physical examination, brain magnetic resonance imaging, FMA-UE, WMFT, modified Ashworth scale, ect.
2. Surgery follow-up timepoint (V2): All participants will be implanted with the VNS system, including the G115R IPG and L312 lead.
3. Baseline follow-up timepoint (V3): There is a baseline evaluation 7 to 14 days after the surgery, then participants will be randomly assigned to VNS group or Control group.
4. Clinic rehabilitation follow-up timepoint (V4): Participants will receive standard clinic rehabilitation 3 days per week and lasting 6 weeks. Both active VNS group (VNS group) and sham VNS group (Control group) will receive rehabilitation. Participants will be evaluated at the last day of this follow-up timepoint.
5. Home exercise follow-up timepoint (V5): Participants will take standard home exercise everyday in 6 weeks. Both active VNS group (VNS group) and sham VNS group (Control group) will receive rehabilitation. At the last day, after evaluating, group assignment is unblinded.
6. Unmasking follow-up timepoint (V6): In this 6 weeks, all participants will receive active VNS. Participants in VNS group will still take standard home exercise, and participants in Control group will receive standard clinic rehabilitation again. Participants will be also evaluated at the last day of this follow-up timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years and <80 years, all gender is acceptable.
* History of unilateral supratentorial intracerebral hemorrhage ≥ 6 months but < 5 years.
* Upper Extremity motor section of the Fugl-Meyer Assessment score ≥20 and ≤50.
* Right- or left-sided weakness of upper extremity.
* Ability to communicate, understand, and give appropriate consent. Subjects can follow trial commands.
* Subjects have good compliance and can complete the visits after surgery.

Exclusion Criteria:

* History of ischemic stroke.
* Cerebral hemorrhage resulting from tumors, trauma, aneurysms, or hemorrhagic transformation of ischemic stroke.
* Presence of ongoing dysphagia or aspiration difficulties.
* Prior injury to vagus nerve, either bilateral or unilateral.
* Subject receiving medication that may significantly interfere with actions of VNS on neurotransmitter systems at study entry, clinic rehabilitation follow-up timepoint, or home rehabilitation follow-up timepoint, such as centrally acting cholinoceptor blockers, centrally acting adrenoceptor blockers, norepinephrine re-uptake inhibitors, etc.
* Botox injections within 4 weeks prior to enrollment through the unmasking follow-up timepoint (Visit 6).
* Severe spasticity of the upper extremity (Modified Ashworth ≥ 3).
* Significant sensory loss of the upper extremity (Upper Extremity sensory section of the Fugl-Meyer Assessment score < 6).
* Current requirement, or likely future requirement, of diathermy.
* Current use of any other stimulation device, such as a pacemaker or other neurostimulator.
* Pregnancy or plans to become pregnant or to breastfeed during the study period.
* Participated in any other clinical trials within the preceding 3 months.
* Not considered to be applicable by the investigator.

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Average Change | V4, 6 weeks after baseline follow-up timepoint
  The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment). The FMA-UE will be analyzed for difference in average change at Clinic rehabilitation follow-up timepoint compared to Baseline follow-up timepoint (Difference in average change in FMA-UE from V3 to V4).

SECONDARY OUTCOMES:
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Response | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint
  The Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Response is the percent of patients with a 6 point or greater improvement on the FMA-UE.
Upper Extremity Motor Section of the Fugl-Meyer Assessment (FMA-UE) Average Change | V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).
Wolf Motor Function Test (WMFT) Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The Wolf Motor Function Test (WMFT) is an assessment scale of upper extremity functional level after stroke. The functional assessment range is an average of 15 sub-items with a range from 0 to 5, with 0 (meaning did not attempt) to 5 (meaning normal).
Wolf Motor Function Test (WMFT) Response | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint
  Wolf Motor Function Test (WMFT) Response is the percent of patients with a 0.4 point or greater improvement on the WMFT.
EQ-5D-3L Average Change | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The EQ-5D-3L is a general measure of health outcomes in any population. It is a self-report questionnaire which provides a simple descriptive profile and a single index value for health status.
Incidence of Adverse Events | V4, 6 weeks after Baseline follow-up timepoint; V5, 6 weeks after Clinic rehabilitation follow-up timepoint; V6, 6 weeks after Home exercise follow-up timepoint
  The incidence of adverse events occurred during the clinical trial, whether or not related to the device.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxin Lin, Principal Investigator — First Affiliated Hospital of Fujian Medical University

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified case data are available from the authors upon reasonable request, after request in writing to the corresponding authors and after approval by the study committee and principal investigators from each site.